CLINICAL TRIAL: NCT00957879
Title: Effect of Different Vitamin D Preparations on Circulating FGF23 Levels in Vitamin D Deficient Caucasian and African-American Men and Women
Brief Title: Different Vitamin D Preparations & FGF23 in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Sherri-Ann M. Burnett-Bowie, Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2009P000567; K23DK073356 (NIH)
Record Dates: First submitted 2009-08-11; First posted 2009-08-13 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D; FGF23; FGF-23; Phosphate
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Ergocalciferols; Calcitriol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ergocalciferol (Active Comparator): Weekly ergocalciferol for 12 weeks
  Interventions: Dietary Supplement: Ergocalciferol
- calcitriol (Active Comparator): Daily calcitriol for 12 weeks
  Interventions: Dietary Supplement: Calcitriol

INTERVENTIONS:
Dietary Supplement: Ergocalciferol — Ergocalciferol 50000 international units by mouth weekly for 12 weeks
  Arms: ergocalciferol
Dietary Supplement: Calcitriol — Calcitriol 0.5 mcg by mouth daily for 12 weeks
  Arms: calcitriol

SUMMARY:
Fibroblast growth factor 23 (FGF23) is a new hormone which controls phosphate and vitamin D levels in humans. Excess FGF23 is associated with an increased risk of death in patients with chronic kidney disease. In this study the investigators are investigating the effects of different forms of vitamin D on FGF23 levels in the blood in order to increase our understanding of how this important hormone works.

DETAILED DESCRIPTION:
Fibroblast growth factor 23 (FGF23) is a novel hormone involved in phosphate and vitamin D physiology. X-linked hypophosphatemia (XLH), autosomal dominant hypophosphatemic rickets (ADHR), and tumor induced osteomalacia (TIO) are 3 rare diseases characterized by rickets/osteomalacia, fractures, and hypophosphatemia secondary to renal phosphate wasting and inappropriately low levels of activated vitamin D (calcitriol), which are caused by excess amounts of or mutated FGF23. FGF23 excess also occurs in renal failure, where elevated FGF23 levels predict increased mortality. Thus, abnormal FGF23 appears to be central to both rare and common diseases. While FGF23 appears to be regulated by vitamin D, dietary and serum phosphate, much is still unknown. The effects of different forms of vitamin D on FGF23 stimulation are not well characterized. Similarly, any racial differences in the regulation of FGF23 by vitamin D have not been investigated.

To address these knowledge deficits, we will randomize 52 vitamin D deficient (25OHD < or = 24 ng/mL by LC/MS) Caucasian and African-American men and women to treatment with either dietary vitamin D or activated vitamin D for 12 weeks. Our primary endpoint will be the change in FGF23 with dietary versus activated vitamin D.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 45 yrs
* Serum 25OHD < 24 ng/mL by liquid chromatography/mass spectroscopy
* At least 1 menses in the last 3 months (females) and normal serum testosterone (males)
* African-American or Caucasian race

Exclusion Criteria:

* Significant cardiac, hepatic, oncologic, or psychiatric disease
* History of malabsorption, kidney stones, or recent alcohol excess/abuse
* Use of medications known to affect serum phosphate levels including phosphate-binding antacids, sodium etidronate, calcitonin, excessive doses of vitamin D (> 1000 units per day), excessive doses of vitamin A (> 20,000 units/day), calcitriol, growth hormone, or anti-convulsants
* Use of thiazide diuretics or cholestyramine
* Serum calcium < 8 or > 11 mg/dL, creatinine > 1.5 mg/dL, or Hgb < 11 gm/dL
* Serum glucose >140mg/dL
* Liver function tests > 2 times the upper limit of normal
* TSH < 0.1 or > 7 uU/mL
* WBC < 2,000 or > 15,000/cmm
* Platelet count < 100,000 or > 500,000/cum
* Hormone replacement therapy (however, oral contraceptives are allowed) or testosterone use
* Urine beta-hCG positive (females)
* Serum phosphate > 4.6 mg/dL
* Allergy to vitamin D

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2009-05; Primary Completion 2010-09 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Change in FGF23 levels | 12 weeks

SECONDARY OUTCOMES:
Change in serum phosphate | 12 weeks
Change in urinary phosphate | 12 weeks
Change in serum calcium | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sherri-Ann M Burnett-Bowie, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Burnett SM, Gunawardene SC, Bringhurst FR, Juppner H, Lee H, Finkelstein JS. Regulation of C-terminal and intact FGF-23 by dietary phosphate in men and women. J Bone Miner Res. 2006 Aug;21(8):1187-96. doi: 10.1359/jbmr.060507. PMID 16869716
- [Background] Bhan I, Shah A, Holmes J, Isakova T, Gutierrez O, Burnett SM, Juppner H, Wolf M. Post-transplant hypophosphatemia: Tertiary 'Hyper-Phosphatoninism'? Kidney Int. 2006 Oct;70(8):1486-94. doi: 10.1038/sj.ki.5001788. Epub 2006 Aug 30. PMID 16941023
- [Background] Burnett-Bowie SM, Mendoza N, Leder BZ. Effects of gonadal steroid withdrawal on serum phosphate and FGF-23 levels in men. Bone. 2007 Apr;40(4):913-8. doi: 10.1016/j.bone.2006.10.016. Epub 2006 Dec 8. PMID 17157573
- [Background] Burnett-Bowie SM, Henao MP, Dere ME, Lee H, Leder BZ. Effects of hPTH(1-34) infusion on circulating serum phosphate, 1,25-dihydroxyvitamin D, and FGF23 levels in healthy men. J Bone Miner Res. 2009 Oct;24(10):1681-5. doi: 10.1359/jbmr.090406. PMID 19419295